CLINICAL TRIAL: NCT04206033
Title: Hemophilia and Bone Metabolism: Study of Monocytic Populations and Inflammatory Proteins
Acronym: BOHEM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0446
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia; Osteopenia; Arthropathy
MeSH Terms: conditions — Hemophilia A; Bone Diseases, Metabolic; Joint Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
The investigators propose, as part of the study, to carry out for each patient:

* An analysis of monocytic populations by flow cytometry (CD14, CD16, CD45, CD68, CD115, CCR2, CX3CR1, CD163 and CD206).
* A population assessment of Myeloid-Derived Suppressor Cells (MDSC).
* Assays of cytokines and chemokines involved in inflammation by multiplex analyzes: Il-1 (α and β), Il-4, Il-6, Il-10, Il-13, TNF- α, TGF- β, CRP , leptin, IFN- β.
* Specialized dosages of proteins involved in bone metabolism. RANKL, osteoprotegerin, M-CSF, TRAPCP5.

ELIGIBILITY:
Inclusion Criteria:

* Major patients followed at the hemophilia treatment reference center,
* Presenting the diagnosis of severe, moderate or minor Hemophilia A / B,
* Having a social security system,
* Obtaining the oral non-objection collection from the patient after information.

Exclusion Criteria:

* Minor patients, under guardianship or curatorship.
* Causes of secondary osteoporosis:

  * Systemic corticosteroid therapy in progress (≥ 3 consecutive months, at a dosage ≥ 7.5 mg / d of prednisone equivalent).
  * other treatment or condition responsible for osteoporosis: prolonged or medicated hypogonadism, untreated active hyperthyroidism, hypercorticism, primary hyperparathyroidism.
* Treatment with biphosphonates, biotherapies or hormone therapy in the treatment of prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will include adult male patients with hemophilia A or B, severe, moderate or minor.
  In addition, the investigators will include patients with Hemophilia A with an inhibitor.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To study the monocytic populations possibly involved in bone metabolism in hemophiliac patients. | 1 year
  Evaluation of the inflammatory profile of patients by protein assays

SECONDARY OUTCOMES:
Find a correlation between the main objective and the measurement of bone density | 1 year
  Evaluation of biochemical parameters involved in bone metabolism
Find a correlation between the main objective and the measurement of bone density | 1 year
  Non-invasive bone mineral density measurement
Look for a correlation between the main objective and physical activity | 1 year
  Assessment of physical activity by self-questionnaire
Look for a correlation between the main objective and the inflammatory profile in hemophiliac patients. | 1 year
  Evaluation of the inflammatory profile of patients by protein assays

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided